CLINICAL TRIAL: NCT04672304
Title: Factors Affecting the Use of Long Term and Permanent Contraceptive Methods; Cross Sectional Study.
Brief Title: Long Term and Permanent Contraceptive
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, University of Jordan
Other Study IDs: JUH
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Contraceptive Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Al-Husban University Naser — filling a questionnaire

SUMMARY:
We will study with the different variables that affect the intention to use long- acting and permanent contraceptive methods among married women in Jordan through a cross sectional study. Self- administered questionnaire will be distributed to aid in data collection.

DETAILED DESCRIPTION:
In this cross-sectional study, self-administered pre-made questionnaires. (https://docs.google.com/forms/d/e/1FAIpQLSdjuuQynIxu0AAmIbKHg0-iyZgTW0m5847JaX0OZrnl7v7v1w/viewform ) will be distributed to married women. (Women of childbearing age). The candidates will be selected according to their age (15-49), marital status (married), and pregnancy status (non-pregnant). The data collected through the questionnaires will then be processed and interpreted in order to understand the variables that affect the use of LACM and permanent contraception methods among Jordanian women.

ELIGIBILITY:
Inclusion Criteria:

* females used or currently using long-term contraception

Exclusion Criteria:

* never users of contraception

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — females using or used contraception
Study Population: women aged 15-49 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1365 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
The use of LACM and permanent contraception methods measure by a questionnaire | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No